CLINICAL TRIAL: NCT01381484
Title: Efficacy and Safety of Topical Argireline in the Treatment of Periorbital Wrinkles
Brief Title: Argireline in Treatment of Periorbital Wrinkles
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mahidol University (Other)
Collaborators: Pacific Health Foundation (Other)
Responsible Party: Department of dermatology, Mahidol university
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Svarothai
Record Dates: First submitted 2011-03-30; First posted 2011-06-27 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2011-03

CONDITIONS: Wrinkles
Keywords: Periorbital wrinkles; Efficacy and safety
MeSH Terms: interventions — acetyl-glutamyl-glutamyl-methionyl-glutaminyl-arginyl-argininamide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (No Intervention): This group received placebo gel and requested to apply periorbital area and over the face for 3 months.
- Study group (Experimental): This group received La Jolie Gel and requested to apply periorbital area and over the face for 3 months.
  Interventions: Drug: 10% Argireline

INTERVENTIONS:
Drug: 10% Argireline — 10% Argireline (La jolie gel®, Pacific health care, Thailand) were instructed to apply the gel over the face and periorbital area twice daily for a period of 3 months.
  Other Names: 10% Argireline (La jolie gel®)
  Arms: Study group

SUMMARY:
The purpose of this study is to determine whether La Jolie gel is effective in the treatment of periorbital wrinkles.

DETAILED DESCRIPTION:
Argireline has mechanism of action that significantly inhibited neurotransmitter release with a potency similar to that of BoNTA. Inhibition of neurotransmitter release was due to the interference of the hexapeptide with the formation and/or stability of SNARE complex. Notably, this peptide did not exhibit in vivo oral toxicity nor primary irritation at high doses. These findings demonstrate that Argireline is a anti-wrinkle peptide that emulates the action of currently used BoNTs.

In vivo study, Topical Argireline 10% is applied on lateral preorbital area twice daily for 30 days. The result demonstrates a significant anti-wrinkle activity by decreased skin wrinkle 30%. These findings demonstrate a significant anti-wrinkle activity for Argireline, in agreement with its in vitro and cellular activities. Topical Argireline represents a bio-safe alternative to BoNTs in anti-wrinkle therapy.

ELIGIBILITY:
Inclusion Criteria:

* healthy woman at 35-45 years old
* Presence of periorbital wrinkles

Exclusion Criteria:

* Pregnancy
* Nursing
* Keloids /scar at periorbital area
* pre-treatment with topical periorbital products within 1 month
* Botulinum toxin A injection,facial plastic surgery within 1 year
* Allergic to active ingredients including acetyl hexapeptide-3 Argireline®, sodium hyaluronate,adenosine,arbutin,fucus vesiculosus)

Ages: 35 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2009-03; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Efficacy | 3 months
  Objective evaluation
  * Noninvasive measurement by skin bioengineering technique e.g. visioscan, corneometer, cutometer
  * Comparative photographic evaluation by certified dermatologists
  Subjective evaluation
  * Patient Self assessment satifaction review

SECONDARY OUTCOMES:
Safety | 3 months
  Number of participants with adverse events Categorized adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Supenya varothai, M.D., Principal Investigator — Department of Dermatology, Faculty of Medicine Siriraj Hospital, Mahidol University
Locations (1):
- Department of dermatology, Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkoknoi, Bangkok, Thailand

REFERENCES:
- [Background] Blanes-Mira C, Clemente J, Jodas G, Gil A, Fernandez-Ballester G, Ponsati B, Gutierrez L, Perez-Paya E, Ferrer-Montiel A. A synthetic hexapeptide (Argireline) with antiwrinkle activity. Int J Cosmet Sci. 2002 Oct;24(5):303-10. doi: 10.1046/j.1467-2494.2002.00153.x. PMID 18498523
- [Background] Tokiwa Y, Kitagawa M, Raku T, Yanagitani S, Yoshino K. Enzymatic synthesis of arbutin undecylenic acid ester and its inhibitory effect on melanin synthesis. Bioorg Med Chem Lett. 2007 Jun 1;17(11):3105-8. doi: 10.1016/j.bmcl.2007.03.039. Epub 2007 Mar 16. PMID 17418566
- [Result] Farage MA, Miller KW, Elsner P, Maibach HI. Intrinsic and extrinsic factors in skin ageing: a review. Int J Cosmet Sci. 2008 Apr;30(2):87-95. doi: 10.1111/j.1468-2494.2007.00415.x. PMID 18377617
- [Result] Klein AW. Complications, adverse reactions, and insights with the use of botulinum toxin. Dermatol Surg. 2003 May;29(5):549-56; discussion 556. doi: 10.1046/j.1524-4725.2003.29129.x. No abstract available. PMID 12752527
- [Result] Brown MB, Jones SA. Hyaluronic acid: a unique topical vehicle for the localized delivery of drugs to the skin. J Eur Acad Dermatol Venereol. 2005 May;19(3):308-18. doi: 10.1111/j.1468-3083.2004.01180.x. PMID 15857456
- [Result] Abella ML. Evaluation of anti-wrinkle efficacy of adenosine-containing products using the FOITS technique. Int J Cosmet Sci. 2006 Dec;28(6):447-51. doi: 10.1111/j.1467-2494.2006.00349.x. PMID 18489289
- [Result] Senni K, Gueniche F, Foucault-Bertaud A, Igondjo-Tchen S, Fioretti F, Colliec-Jouault S, Durand P, Guezennec J, Godeau G, Letourneur D. Fucoidan a sulfated polysaccharide from brown algae is a potent modulator of connective tissue proteolysis. Arch Biochem Biophys. 2006 Jan 1;445(1):56-64. doi: 10.1016/j.abb.2005.11.001. Epub 2005 Nov 28. PMID 16364234
- [Result] Narins RS, Brandt F, Leyden J, Lorenc ZP, Rubin M, Smith S. A randomized, double-blind, multicenter comparison of the efficacy and tolerability of Restylane versus Zyplast for the correction of nasolabial folds. Dermatol Surg. 2003 Jun;29(6):588-95. doi: 10.1046/j.1524-4725.2003.29150.x. PMID 12786700
- [Result] Rohrich RJ. The increasing popularity of cosmetic surgery procedures: a look at statistics in plastic surgery. Plast Reconstr Surg. 2000 Nov;106(6):1363-5. doi: 10.1097/00006534-200011000-00023. No abstract available. PMID 11083570
- [Result] Manaloto RM, Alster TS. Periorbital rejuvenation: a review of dermatologic treatments. Dermatol Surg. 1999 Jan;25(1):1-9. doi: 10.1046/j.1524-4725.1999.08049.x. PMID 9935084